CLINICAL TRIAL: NCT03241225
Title: EM/PROTECT: Improving Depression in Elder Mistreatment Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York City Department for the Aging (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1703018101; P50MH113838 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Depression
Keywords: Elder abuse; Depression; Mental health
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will compare the effectiveness and target engagement of EM/PROTECT with EM enriched with training of EM staff in linking EM victims to mental health services (EM/MH) in order to position us for a fully powered R01. To ensure rigor and reproducibility, EM/PROTECT or EM/MH will be offered to randomly assigned depressed EM victims, and standard assessments will be conducted by trained raters blind to participant assignment and our hypotheses.
Who Masked: Outcomes Assessor
Masking Description: Standardized assessments will be conducted by trained raters blind to participant assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EM/PROTECT (Experimental): This group of participants will receive the EM/PROTECT intervention, a behavioral intervention for depressed elder mistreatment (EM) victims designed to work in synergy with EM mistreatment resolution services that provide safety planning, support services, and links to legal services.
  Interventions: Behavioral: EM/PROTECT
- EM/MH (Active Comparator): This group of participants experiencing elder mistreatment will receive support services from staff trained in linking elder mistreatment victims to community mental health services.
  Interventions: Behavioral: EM/MH

INTERVENTIONS:
Behavioral: EM/PROTECT — EM/PROTECT is a behavioral intervention for depressed elder mistreatment (EM) victims designed to work in synergy with EM mistreatment resolution services that provide safety planning, support services, and links to legal services
  Arms: EM/PROTECT
Behavioral: EM/MH — EM/MH provides individuals experiencing elder mistreatment with support services from staff trained in linking elder mistreatment victims to community mental health services.
  Arms: EM/MH

SUMMARY:
The investigators developed EM/PROTECT, a behavioral intervention for depressed EM (elderly mistreatment) victims, to work in synergy with EM mistreatment resolution services that provide safety planning, support services, and links to legal services. PROTECT is built on a model which postulates that chronic stress promotes dysfunction of the cognitive control (CCN) and reward networks, impairing the victims' ability to flexibly respond to the environment and limits their reward activities. PROTECT therapists work with victims to develop action plans to reduce stress, and to increase rewarding experiences. EM/PROTECT has been designed in an iterative process with community EM providers of the New York City (NYC) Department for the Aging (DFTA) to use agencies' routine PHQ-9 depression screening and referral for service. In the current study, the investigators will compare the effectiveness of EM/PROTECT with EM enriched with staff training in linking EM victims to community mental health services (EM/MH). The investigators intend to enroll 80 subjects that will participate in the study for approximately 12 weeks.

DETAILED DESCRIPTION:
One in ten older adults is a victim of mistreatment, and one third of victims have clinically significant depressive symptoms. Depression increases mortality and decreases motivation to take self-protective steps. Yet, no elder mistreatment (EM) agencies have embedded identification and treatment of depressed EM victims in their programs. The investigators developed EM/PROTECT, a behavioral intervention for depressed EM victims, to work in synergy with EM agencies that provide safety planning and links to legal services. EM/PROTECT has been designed in an iterative process with community EM providers of the NYC Department for the Aging (DFTA), to utilize agencies' routine depression screening and service referrals. The investigators propose to collect data on the feasibility and acceptability of EM/PROTECT as one of three developmental projects under the ALACRITY Center NIMH grant (1 P50 MH113838-01,PI: Alexopoulos) (IRB 1704018108). We will compare the effectiveness of EM/PROTECT with EM enriched with staff training in linking EM victims to community mental health services (EM/MH). To ensure rigor and reproducibility, EM/PROTECT or EM/MH will be offered to randomly assigned depressed EM victims. All EM victims will receive standard EM resolution services from DFTA. EM staff will screen and refer depressed victims to Cornell staff, who will describe the study and obtain consent. Standardized assessments will be conducted by trained raters blind to participant assignment.

In addition, the investigators will use both active and passive sensing technology through smartphone data collection to supplement in-person data collection with an objective measure of socialization and behavioral activation. Smartphone data will be used to explore whether adherence to active recordings and time spent carrying the phone is associated with greater effectiveness of EM/PROTECT.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Capacity to consent (per EM staff)
* Significant depression (per EM staff) as indicated by a score of 10 or above on the Patient Health Questionnaire-9 (PHQ-9), a widely used screening tool routinely administered in EM agency settings (the PHQ-9 has a sensitivity of 88% and a specificity of 88% for major depression)
* Need for EM services

Exclusion Criteria:

* Active suicidal ideation (MADRS item 10>4)
* Inability to speak English
* Axis 1 DSM-5 diagnoses other than unipolar depression or generalized anxiety disorder (by SCID)
* Mini-Mental Exam score of 23 or less 5
* Severe or life-threatening medical illness
* EM emergency and or referral out of EM agency (per EM staff)

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, MD, Study Director — Weill Cornell Medicine/New York Presbyterian Hospital; Jo Anne Sirey, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Elderly Crime Victim Resource Center of the New York City Department for the Aging, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Center will share its data via the NIMH Data Archive (NDA). Our resource sharing plan is formulated in accordance with the NDA Data Sharing Terms and Conditions. Further, the Center will use NDA technologies to submit data in accordance with the NDA Data Sharing Terms and Conditions. This project will share feasibility, acceptability, and preliminary effectiveness data of the developmental study of the behavioral intervention EM/PROTECT. Investigators will comply with NIMH's procedures for data deposition into NDCT, and will let NDCT policies dictate the timetable upon which and avenues through which others will be allowed to access those data. Investigators will make the dataset available to other researchers after the main results have been published. Investigators will de-identify the data in the final datasets prior to release for sharing.
Time Frame: Per NIMH guidelines
Access Criteria: To ensure data and participant security, investigators will make the data available to users only under a data-sharing agreement. All users will first provide to the ALACRITY Center and the co-Investigators with a proposal of hypotheses, variables needed to test these hypotheses, and plans for dissemination of findings. All users will indicate in a signed document: (1) a commitment to using the data only for research purposes; (2) a plan for securing the data; (3) an agreement to either destroying or returning the data once analyses are completed; and (4) an agreement to not share data with other users and to direct all such requests to The ALACRITY Center.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EM/PROTECT | EM/MH
Started | 24 | 16
Completed | 17 | 14
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EM/PROTECT | EM/MH | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.04 (8.48) | 73.5 (7.53) | 72.77 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 13 | 3 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Clinically Significant Depressive Symptoms (MADRS) [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale. Scores on this scale range from 0 to 60, with higher scores indicating more severe depression and lower scores indicating milder depression.
  units on a scale | 24.21 (3.09) | 22.94 (5.35) | 23.58 (4.22)
Assessment of Quality of Life (WHO-QOL) [Mean (Standard Deviation); unit: units on a scale] — World Health Organization-Quality Of Life scale. The overall scores range between 26-130. In all domains, higher scores indicate better health. Domain 1 measures general health (scores range from 2-10). Domain 2 measures physical health (scores range from 7-35). Domain 3 measures psychological health (scores range from 6-30). Domain 4 measures social health (scores range from 3--15). Domain 5 measures environmental health (scores range from 8-40).
  units on a scale
    Domain 1 | 5.71 (2.27) | 5.44 (2.03) | 5.58 (4.3)
    Domain 2 | 19.33 (5.16) | 20.13 (3.36) | 19.73 (4.26)
    Domain 3 | 18.22 (5.18) | 18.06 (4.04) | 18.14 (4.61)
    Domain 4 | 6.71 (3.01) | 8.44 (2.00) | 7.58 (2.51)
    Domain 5 | 23.58 (7.71) | 23.88 (5.57) | 23.73 (6.64)
Satisfaction With Study Intervention (CSQ) [Mean (Standard Deviation); unit: units on a scale] — Client Satisfaction Questionnaire. Overall scores range from 3-12. Domain 1 measures met needs. Scores range from 1-4 and higher scores indicate more needs met. Domain 2 measures satisfaction with services. Scores range from 1-4 and higher scores indicate more satisfaction with services. Domain 3 measures willingness to return. Scores range from 1-4 and higher scores indicate greater willingness to return.
  units on a scale
    Domain 1 | 2.95 (1.23) | 2.7 (1.49) | 2.83 (1.36)
    Domain 2 | 2.95 (1.23) | 3.00 (1.41) | 2.98 (2.64)
    Domain 3 | 3.30 (1.22) | 3.20 (1.32) | 3.25 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Depressive Symptoms (MADRS).
Description: In both conditions, the reduction of clinically significant depressive symptoms as measured on the Montgomery Asberg Depression Rating Scale (MADRS). Scores on this scale range from 0 to 60, with higher scores indicating more severe depression and lower scores indicating milder depression.
Time Frame: These measures are assessed at baseline, six week, nine week and twelve weeks after study enrollment during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EM/PROTECT | EM/MH
Number analyzed (Participants) | 24 | 16
score on a scale
  Baseline Outcomes | 24.21 (5.35) | 22.94 (3.09)
  Week 6 Outcomes | 12.59 (7.02) | 17.54 (7.21)
  Week 9 Outcomes | 15.80 (5.76) | 22.82 (7.95)
  Week 12 Outcomes | 16.64 (7.87) | 13.05 (7.39)
Statistical Analysis 1: Comparison: EM/PROTECT vs EM/MH; Week 12; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = 3.59, 95% CI 2-sided [-1.43 to 8.61] — Mean change in EM/PROTECT group not significantly different from mean change in EM/MH group, at week 12

2. Secondary Outcome: Assessment of Quality of Life (WHO-QOL)
Description: IN both conditions, improvement in assessment of quality of life measured by the World Health Organization Quality of Life (WHOQOL) scale. The overall scores range between 26-130. In all domains, higher scores indicate better health. Domain 1 measures general health (scores range from 2-10). Domain 2 measures physical health (scores range from 7-35). Domain 3 measures psychological health (scores range from 6-30). Domain 4 measures social health (scores range from 3--15). Domain 5 measures environmental health (scores range from 8-40).
Time Frame: These measures are assessed at baseline, six week, nine week and twelve weeks after study enrollment during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EM/PROTECT | EM/MH
Number analyzed (Participants) | 24 | 16
score on a scale
  Domain 1- Baseline | 5.71 (2.27) | 5.44 (2.03)
  Domain 2- Baseline | 19.33 (5.16) | 20.13 (3.36)
  Domain 3- Baseline | 18.22 (5.18) | 18.06 (4.04)
  Domain 4- Baseline | 6.71 (3.01) | 8.44 (2.00)
  Domain 5- Baseline | 23.58 (7.71) | 23.88 (5.57)
  Domain 1- Week 6 | 6.70 (1.81) | 4.83 (3.04)
  Domain 2- Week 6 | 21.30 (3.33) | 16.17 (7.99)
  Domain 3- Week 6 | 19.30 (4.23) | 16.90 (3.41)
  Domain 4- Week 6 | 5.20 (2.09) | 6.42 (3.55)
  Domain 5- Week 6 | 26.85 (5.76) | 19.92 (10.56)
  Domain 1- Week 9 | 5.93 (2.64) | 6.82 (1.70)
  Domain 2- Week 9 | 20.14 (7.15) | 22.59 (2.87)
  Domain 3- Week 9 | 18.62 (4.23) | 19.53 (4.90)
  Domain 4- Week 9 | 8.64 (3.37) | 7.94 (2.11)
  Domain 5- Week 9 | 23.79 (8.32) | 27.00 (5.28)
  Domain 1- Week 12 | 6.41 (2.00) | 6.57 (1.74)
  Domain 2- Week 12 | 21.88 (3.16) | 20.50 (3.18)
  Domain 3-Week 12 | 20.47 (4.29) | 25.00 (19.43)
  Domain 4- Week 12 | 7.76 (1.99) | 13.00 (8.36)
  Domain 5- Week 12 | 26.59 (3.02) | 27.21 (5.01)
Statistical Analysis 1: Comparison: EM/PROTECT vs EM/MH; Domain #1, Week 12; Test type: Superiority; p = 0.79, t-test, 2 sided; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-1.37 to 1.05]
Statistical Analysis 2: Comparison: EM/PROTECT vs EM/MH; Domain #2, Week 12; Test type: Superiority; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-0.70 to 3.46]
Statistical Analysis 3: Comparison: EM/PROTECT vs EM/MH; Domain #3, Week 12; Test type: Superiority; p = 0.37, t-test, 2 sided; Mean Difference (Final Values) = -4.53, 95% CI 2-sided [-14.99 to 5.93]
Statistical Analysis 4: Comparison: EM/PROTECT vs EM/MH; Domain #4, Week 12; Test type: Superiority; p = 0.026, t-test, 2 sided; Mean Difference (Final Values) = -5.24, 95% CI 2-sided [-9.75 to -0.73]
Statistical Analysis 5: Comparison: EM/PROTECT vs EM/MH; Domain #5, Week 12; Test type: Superiority; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-3.51 to 2.27]

3. Other Pre Specified Outcome: Satisfaction With Study Intervention (CSQ)
Description: Client satisfaction with study intervention as measured by the Client Satisfaction Questionnaire (CSQ) in both treatments. Overall scores range from 3-12. Domain 1 measures met needs. Scores range from 1-4 and higher scores indicate more needs met. Domain 2 measures satisfaction with services. Scores range from 1-4 and higher scores indicate more satisfaction with services. Domain 3 measures willingness to return. Scores range from 1-4 and higher scores indicate greater willingness to return.
Time Frame: Assessed after EM/PROTECT sessions completed at six, nine, and twelve weeks after study enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EM/PROTECT | EM/MH
Number analyzed (Participants) | 24 | 16
score on a scale
  Domain 1- Week 6 | 2.95 (1.2) | 2.70 (1.49)
  Domain 2- Week 6 | 2.95 (1.23) | 3.00 (1.41)
  Domain 3- Week 6 | 3.30 (1.22) | 3.20 (1.32)
  Domain 1- Week 9 | 3.00 (1.06) | 2.31 (1.70)
  Domain 2- Week 9 | 3.29 (1.05) | 2.69 (1.89)
  Domain 3- Week 9 | 3.41 (1.00) | 2.54 (1.81)
  Domain 1- Week 12 | 3.12 (0.93) | 2.42 (1.68)
  Domain 2- Week 12 | 3.53 (0.62) | 2.75 (1.71)
  Domain 3- Week 12 | 3.65 (0.61) | 3.00 (1.81)
Statistical Analysis 1: Comparison: EM/PROTECT vs EM/MH; Domain #1, Week 12; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-0.26 to 1.66]
Statistical Analysis 2: Comparison: EM/PROTECT vs EM/MH; Domain #2, Week 12; Test type: Superiority; p = 0.047, t-test, 2 sided — Domain #2; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [0.011 to 1.55]
Statistical Analysis 3: Comparison: EM/PROTECT vs EM/MH; Domain #3, Week 12; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.34 to 1.64]

ADVERSE EVENTS:
Time Frame: Assessed at 6 weeks, 9 weeks, and 12 weeks after study enrollment.
Arm/Group | EM/PROTECT | EM/MH
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/16
Serious Adverse Events (participants affected / at risk) | 3/24 | 3/16
Other Adverse Events (participants affected / at risk) | 0/24 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EM/PROTECT (N=24) | EM/MH (N=16)
Dehydration (General disorders) | 1 (1) | 0 (0) — Participant visited the emergency room due to dehydration.
Stomach surgery (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant had a planned surgery to remove a stomach mass
Loss of consciousness (General disorders) | 1 (1) | 0 (0) — Participant lost consciousness during a planned doctor's visit
Heart attack (Cardiac disorders) | 0 (0) | 1 (1) — Participant suffered a heart attack
Pneumonia (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Participant diagnosed with pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EM/PROTECT (N=24) | EM/MH (N=16)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant fell in their home

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT03241225/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT03241225/SAP_001.pdf